CLINICAL TRIAL: NCT04536064
Title: COMBINATION OF LYMPHATICO-VENULAR ANASTOMOSIS AND LIPOSUCTION TO TREAT CANCER-RELATED LYMPHEDEMA: RATIONALE FOR A REGIONAL APPROACH
Brief Title: COMBINATION OF LYMPHATICO-VENULAR ANASTOMOSIS AND LIPOSUCTION IN TREATING LYMPHEDEMA
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Siena (Other)
Responsible Party: Principal Investigator, Guido Gabriele, MD, University of Siena
Other Study IDs: LVA+LIPOSUCTION IN LYMPHEDEMA
Record Dates: First submitted 2020-08-27; First posted 2020-09-02 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Description of an Effective Surgical Strategy to Treat Cancer Related Lymphedema, a High Incidence Pathology
Keywords: lymphedema; lva; liposuction; treatment
MeSH Terms: conditions — Lymphedema | interventions — Lipectomy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: LVA and liposuction — Tumescent technique in lymph-sparing fashion was adopted. Areas were infiltrated with a mix of a standard tumescent solution consisting for each liter of in 1000 ml of saline solution, 50 ml lidocaine 1%, 1 ml epinephrine 1:1000, 10 ml bicarbonate 8,4%. Infiltration volume was approximately from 0,5 to 1 liter for the upper extremities and 1-2 liters for lowers. Three to 4 mm 3 holes blunt cannulas were employed. Aspiration technique was as parallel as possible along the lymphatic network pattern and from superficial to deep layers.
  Lymphatic vessels identified at ICG lymphography were spared. Volume of the aspirate was aimed to approximate 80 percent of the volume difference between the affected and non affected side.
  The number and type of anastomosis were recorded as well as amount of removed lipoaspirate versus the excess limb volume.

SUMMARY:
* cooperation of an International team with many years of experience in surgical management of lymphedema
* description of an effective surgical strategy to treat cancer-related lymphedema, a high incidence pathology
* the combination of LVA and liposuction guarantees long lasting results

DETAILED DESCRIPTION:
Cancer-related lymphedema represents one of the major complications of cancer treatment, especially for breast and gynecologic cancers. Moreover, it has high impact on cancer survivors and healthcare systems. Lymphedema management still remains challenging. The better understanding of lymphedema physiopathology as well as the development of sophisticated surgical and diagnostic techniques have led to effective strategies to address lymphedema patients but, despite the considerable interest in international literature, no consensus exist.

The authors present a retrospective analysis of 24 consecutive patients affected by cancer-related lymphedema treated by the combination of LVA and liposuction in the same surgical session. Patients data regarding limb volume, lymphangitis rate and quality of life index were assessed before surgery and 1 year after surgery.

One year after surgery an average volume reduction of 37,9% was registered. Lymphangitis rate significantly decreased after surgery to 0.95 per year. Quality of life score improved.

CONCLUSIONS The combination of LVA and liposuction represents an effective strategy in treating patients with cancer-related lymphedema, ensuring a significant decrease in volume and reduction of lymphangitis rate as well as stable results in time. In addition, it appears to be minimally invasive and well tolerated by patients, since it can be performed under local anesthesia with low risk of complications.

ELIGIBILITY:
Inclusion Criteria:

previous lymphadenectomy

Exclusion Criteria:

free from cancer related pathology

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: 24 patients with secondary lymphedema
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Volume reduction of the limb | one year after surgery
  mesurement of volume reduction

CONTACTS AND LOCATIONS:
Locations (1):
- Guido Gabriele, Siena, SI, Italy

IPD SHARING:
Plan to Share IPD: Undecided